CLINICAL TRIAL: NCT06030765
Title: Evaluation of Rapid Cognitive Screening Tools for Detection of Cognitive Impairment in Older Surgical Patients: A Prospective Cohort Study - Detect CI Study
Brief Title: Detect CI (Cognitive Impairment) Study
Acronym: CI
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5810
Record Dates: First submitted 2023-08-11; First posted 2023-09-11 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Impairment (CI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective multicenter cohort study which will evaluate rapid (administration time ≤ 5 minutes) cognitive screening tools that can be administered preoperatively in older patients undergoing noncardiac surgery. Namely, our study will determine the diagnostic accuracy (sensitivity, specificity, and area under the curves [AUC]) of two rapid, easily administered cognitive screening tools: the Mini-Cog and the Ascertain Dementia 8-item Questionnaire (AD8) against the Montreal Cognitive Assessment (MoCA). Additionally, we will examine the prevalence of cognitive impairment (CI) in patients meeting the CI criteria by either the AD8, Mini-Cog, MoCA, or a single cognitive question from the Centers for Disease Control and Prevention [CDC]. This study will target older patients from surgical offices and/or pre-admission clinics at Toronto General (TGH), Toronto Western (TWH), and Mount Sinai Hospital (MSH), Toronto, Ontario. The identification and recruitment of eligible patients will be a collaborative effort between the nurses, surgeons, anesthesiologists, and the research team. Written informed consent to participate in the study will be obtained from all patients.

DETAILED DESCRIPTION:
The primary aims of the study is to (1) determine the diagnostic accuracy (sensitivity, specificity, and the AUC) of two rapid cognitive screening tools (AD8 and Mini-Cog) against the MoCA in the older surgical population and (2) determine the prevalence of CI as detected by the cognitive screening tests (AD8, Mini-Cog, MoCA, or CDC cognitive question). The secondary aims are to (1) compare the trajectory of patient-reported outcomes at baseline, 30-, and 90-day post-surgery in patients with or without CI as detected by the cognitive screening tests, and (2) compare clinical outcomes in patients with or without CI as detected by the cognitive screening tests.

The study consists of four consecutive time points, including one preoperative assessment and three postoperative assessments occurring during participants' hospital stay and at 30- and 90-day post-surgery. In the preoperative assessment 1-30 days before their scheduled surgery, patients will be asked to complete the AD8, Mini-Cog, MoCA, CDC cognitive question, and the STOP-Bang Questionnaire in-person.

Additionally, patients will be asked to complete the following assessments via an online survey, over the telephone, or in-person prior to their scheduled surgery: WHODAS-2.0 (World Health Organization Disability Assessment Schedule 2.0), 5-item FRAIL Questionnaire, PHQ-4 (4-Item Patient Health Questionnaire for Anxiety and depression), VAS (visual analog scale) pain, SQS (Single Item Sleep Quality Scale), and a single question on QoL (quality of life).

The first postoperative time point will occur during participants' stay at the hospital in which postoperative delirium (POD), postoperative complications, length of stay (LOS), and discharge destination will be assessed. At 30- and 90-day postoperatively, chart review will be performed to assess clinical outcomes, such as postoperative complications, all-cause mortality, and hospital readmission. Patient-reported outcomes, including WHODAS 2.0, 5-item FRAIL Questionnaire, PHQ-4, VAS pain, and QoL, will also be assessed through an online survey or over the telephone.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 65 years old;
* competent to provide informed consent in English;
* undergoing elective non-cardiac surgery;
* education ≥ 8 years;
* able to be contacted by telephone.

Exclusion Criteria:

* previous neurocognitive disorder (e.g., dementia) diagnosis;
* uncontrolled psychiatric disorders;
* hearing and/or vision impairment;
* unable to write or hold pen;
* undergoing neurosurgery;
* unable to provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients scheduled to undergo elective inpatient non-cardiac surgery under general and/ or regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy (sensitivity, specificity | Pre-surgery
  The diagnostic accuracy (sensitivity and specificity) of the AD8 (Eight-item Interview to Differentiate Aging and Dementia) and Mini-Cog against the MoCA (Montreal Cognitive Assessment).
The diagnostic accuracy (AUC) | Pre-surgery
  The AUC (Area under the Receiver Operating Characteristic Curve (ROC)) of the AD8 (Eight-item Interview to Differentiate Aging and Dementia) and Mini-Cog against the MoCA (Montreal Cognitive Assessment).
Prevalence of cognitive impairment (CI) via cognitive screening tools | Pre-surgery
  The prevalence of CI as detected by the AD8 (Eight-item Interview to Differentiate Aging and Dementia). The AD8 is scored from 0-8 with a score of two or more indicating cognitive impairment.
Prevalence of cognitive impairment (CI) via cognitive screening tools | Pre-surgery
  The prevalence of CI as detected by the Mini-Cog. The Mini-Cog is scored from 0-5 with a score of two or less indicating cognitive impairment.
Prevalence of cognitive impairment (CI) via cognitive screening tools | Pre-surgery
  The prevalence of CI as detected by the MoCA (Montreal Cognitive Assessment). The MoCA is scored from 0-30 with a score of 25 or less indicating cognitive impairment.
Prevalence of cognitive impairment (CI) via cognitive screening tools | Pre-surgery
  The prevalence of CI as detected by the CDC (Centers of Disease Control and Prevention) cognitive question. The CDC cognitive question is a simple yes or no question, with a response of yes indicating cognitive impairment.

SECONDARY OUTCOMES:
Trajectories and prevalence or incidence of patient-reported outcomes pre-surgery | Pre-surgery, 30- and 90-days post-surgery
  The trajectory and prevalence or incidence of functional disability as measured through the WHODAS 2.0 (World Health Organization Disability Assessment Schedule 2.0) in participants with CI vs those without. A five-point rating scale is used for each question (none = 0, mild = 1, moderate = 2, severe = 3, extreme/cannot do = 4), and a higher WHODAS score indicates greater disability.
Trajectories and prevalence or incidence of patient-reported outcomes pre-surgery | Pre-surgery, 30- and 90-days post-surgery
  The trajectory and prevalence or incidence of frailty as measured through the 5-item FRAIL questionnaire in participants with CI vs those without. It is scored from 0-5 where higher scores indicate frailty.
Trajectories and prevalence or incidence of patient-reported outcomes pre-surgery | Pre-surgery, 30- and 90-days post-surgery
  The trajectory and prevalence or incidence of pain as measured through the VAS Pain (Visual Analog Scale for Pain) in participants with CI vs those without. It is scored from 0-10 where a lower score indicates worse pain.
Trajectories and prevalence or incidence of patient-reported outcomes pre-surgery | Pre-surgery, 30- and 90-days post-surgery
  The trajectory and prevalence or incidence of depression and anxiety as measured through the PHQ-4 (4-Item Patient Health Questionnaire) in participants with CI vs those without. It is scored from 0-12 where a higher score indicates depression and anxiety.
Trajectories and prevalence or incidence of patient-reported outcomes pre-surgery | Pre-surgery
  The trajectory and prevalence or incidence of obstructive sleep apnea (OSA) as measured through the STOP-Bang Questionnaire in participants with CI vs those without. It is scored from 0-8 where a higher score indicates higher risk for OSA.
Trajectories and prevalence or incidence of patient-reported outcomes pre-surgery | Pre-surgery
  The trajectory and prevalence or incidence of sleep disturbances as measured through the SQS (Single Item Sleep Quality Scale) in participants with CI vs those without. It is scored from 0-10 where a lower score indicates sleep disturbances.
Trajectories and prevalence or incidence of patient-reported outcomes pre-surgery | Pre-surgery, 30- and 90-days post-surgery
  The trajectory and prevalence or incidence of quality of life as measured through the single question on Quality of Life (QoL) in participants with CI vs those without. It is scored from 0-100 where a lower score indicates worse quality of life.
Incidence of clinical outcomes post-surgery | 1-3 days post-surgery
  Incidence of postoperative delirium as assessed by the Confusion Assessment Method (CAM) conducted by the nursing team and through medical chart review.
Incidence of adverse clinical outcomes post-surgery | 1-3 days post-surgery
  Incidence of postoperative complications
Clinical outcomes post-surgery | 1-3 days post-surgery
  Hospital length of stay (LOS)
Clinical outcomes post-surgery | 1-3 days post-surgery
  Discharge destination (assess where the participant will be discharged to once out of hospital up to 30-days post-op)
Incidence of adverse clinical outcomes post-surgery | 30- and 90-days post-surgery
  Incidence of mortality
Incidence of adverse clinical outcomes post-surgery | 30- and 90-days post-surgery
  Incidence of readmission
Incidence of adverse clinical outcomes post-surgery | 30- and 90-days post-surgery
  Incidence of postoperative complications
Incidence of adverse clinical outcomes post-surgery | 30- and 90-days post-surgery
  Incidence of emergency department visit
Incidence of adverse clinical outcomes post-surgery | 30- and 90-days post-surgery
  Incidence of re-operation or revision surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - 399 Bathurst St., Toronto Western Hospital, Dept. of Anesthesia, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario